CLINICAL TRIAL: NCT01067859
Title: A Placebo Controlled, Randomized, Double-Blind, Fixed-dose, Multicenter, Phase IIb Study to Investigate the Efficacy and Tolerability of Low Dose BAY58-2667 (25 µg/h, 10 µg/h) Given Intravenously to Subjects With Acute Decompensated Chronic Congestive Heart Failure (ADHF)
Brief Title: A Phase IIb Study to Investigate the Efficacy and Tolerability of Lower Doses Cinaciguat (25 µg/h, 10 µg/h) Given Intravenously to Patients With Acute Decompensated Chronic Congestive Heart Failure (ADHF)
Acronym: COMPOSE 2
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14663; 2009-014378-16 (EudraCT Number)
Record Dates: First submitted 2010-02-11; First posted 2010-02-12 (Estimated); Last update posted 2015-10-08 (Estimated); Status verified 2014-11

CONDITIONS: Acute Heart Failure
Keywords: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — BAY 58-2667

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm 1 (Experimental)
  Interventions: Drug: Cinaciguat (BAY58-2667)
- Arm 2 (Experimental)
  Interventions: Drug: Cinaciguat (BAY58-2667)
- Arm 3 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cinaciguat (BAY58-2667) — Infusion of 25 µg/h during 48 hours
  Arms: Arm 1
Drug: Cinaciguat (BAY58-2667) — Infusion of 10 µg/h during 48 hours
  Arms: Arm 2
Drug: Placebo — Infusion of placebo during 48 hours
  Arms: Arm 3

SUMMARY:
A placebo controlled, double-blind and randomized study to assess different doses of a new drug (BAY58-2667) given intravenously, to evaluate if it is safe and can help to improve the well-being of patients with acute decompensated heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Male and non-pregnant, non-lactating female subjects, age >/= 18 years of age; or women without childbearing potential defined as postmenopausal women aged 55 years or older, women with bilateral tubal ligation, women with bilateral ovariectomy, and women with a hysterectomy
* Subjects must have the clinical diagnosis of Congestive Heart Failure (CHF) made at least three months prior to enrollment
* Subjects must experience worsening of both of the symptoms below leading to hospitalization at the time of entry into the study:

  * dyspnea and
  * clinical evidence of volume overload

Exclusion Criteria:

* Acute de-novo heart failure
* Acute myocardial infarction and/or myocardial infarction within 30 days
* Valvular heart disease requiring surgical intervention during the course of the study
* Heart failure due to or associated with uncorrected primary valvular disease, malfunctioning artificial heart valve, or uncorrected congenital heart disease
* Primary hypertrophic cardiomyopathy
* Acute inflammatory heart disease, eg, acute myocarditis
* Unstable angina requiring angiography

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2010-03; Primary Completion 2010-09 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Pulmonary Capillary Wedge Pressure | 8 hours

SECONDARY OUTCOMES:
Cardiac index (CI) | 8 hours and 48 hours
Kansas City Cardiomyopathy Questionnaire (KCCQ) | Follow up (after 30+5 days)
Right atrial pressure (RAP) | 8 hours and 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (26):
- United States (6):
  - Birmingham, Alabama
  - Jacksonville, Florida
  - Boston, Massachusetts
  - Cincinnati, Ohio
  - Columbus, Ohio
  - Philadelphia, Pennsylvania
- Argentina (2):
  - Quilmes, Buenos Aires
  - Buenos Aires, Ciudad Auton. de Buenos Aires
- Austria (2):
  - Graz, Styria
  - Innsbruck, Tyrol
- Belgium (3):
  - Aalst
  - Bruxelles - Brussel
  - Leuven
- France (3):
  - Créteil
  - Paris
  - Toulouse
- Germany (5):
  - Bad Krozingen, Baden-Wurttemberg
  - Bad Nauheim, Hesse
  - Bad Oeynhausen, North Rhine-Westphalia
  - Düsseldorf, North Rhine-Westphalia
  - Berlin, State of Berlin
- Dublin, Ireland
- Mexico (3):
  - Guadalajara, Jalisco
  - Mexico City, Mexico City
  - México D.F.
- Quezon City, Philippines

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/